CLINICAL TRIAL: NCT04789083
Title: The Effect of Propolis in Tinea Pedis Treatment: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Rukiye Burucu, Assit. Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NecmettinErbakanU-Burucu
Record Dates: First submitted 2020-12-10; First posted 2021-03-09 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Nurse's Role; Patient Education; Foot Care
Keywords: nursing; nurse coaching; patient education; complementary therapy; althernative therapy

STUDY DESIGN:
Intervention Model Description: This study is a double blind randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Propolis) (Experimental): Medical therapy and propolis
  Interventions: Other: Propholis extrate
- Group 2 (Nurse Coaching/ Nursing education) (Experimental): Medical treatment and nurse coaching
  Interventions: Other: Propholis extrate
- Group 3 (Plassebo) (Placebo Comparator): Medical treatment and plassebo will be applied.
  Interventions: Other: Propholis extrate

INTERVENTIONS:
Other: Propholis extrate — Plassebo
  Other Names: Nurse coaching/ Nursing education

SUMMARY:
Tineapedis is an important health problem. Providing foot care in tinea pedis treatment contributes positively to the treatment. In addition, alternative treatments can also be used. In this study, the randomization study group will be divided into three. Medical treatment and foot care training will be applied to the first group, medical treatment and propolis to the second group, medical treatment and plassebo to the control group. Foot care training will be given by nurse coaching. Times of all three groups and their response to treatment will be evaluated.

DETAILED DESCRIPTION:
1. Study Identification: Randomised Controlled Trial
2. Study Status: This will begin
3. Sponsor/Collaborators: SBS Scientific Bio Solutions Inc.
4. Oversight: Patients will be given foot care training. At the same time, a phone call will be provided by the research nurse every week. Evaluation will be made at the end of 2 months
5. Study Description

   It was planned as a double-blind randomized controlled study. The person conducting the randomizer, the person making the statistics and the person performing the medical examiner will be blinded. Power analysis was made using the G * Power (3.1.9.4) program, 0.05 margin of error and 85% power were accepted. A total of 96 people were divided into three groups. Groups were composed of 36 people, including 10% losses for each group.

   Inclusion Criteria:

   Not being pregnant Not being breastfeeding Not having confusion Not being immunosuppressed Not using systemic cortisone Not having any dermatological problems (psoriasis, contact dermatitis, etc.) that will affect the treatment.

   Agree to participate in research Being accessible by phone Having no problems communicating by phone Not having problems with physical care

   Exclusion Criteria:

   Pregnant / nursing women Using systemic antifungal therapy Using systemic croticosteroids In the process of treatment for oncological reasons Are using immunosuppressants Dermatological disease (contact dermatitis, psoriasis) Under the age of 18 and over the age of 64 Have cognitive problems There is no telephone / telephone number within reach Individuals who have difficulties in speaking and understanding Turkish will be excluded from the study.

   Medical treatment applied to all three groups: Sertaconazole nitrate (2%), 1x1, externally Terbinafine hydrochloride (250 mg), 1x1, oral Propolis treatment: Alcoholic extract of propolis will be used topically 2x1. Plassebe: Sterile distilled water 2x1 will be used. Plassebo and propolis extrat will be prepared in the same packages.

   Nurse coaching will continue by the nurse, who received coaching training, using the training booklet, with the first meeting face-to-face and subsequent calls over the phone. Interviews will be held once every two weeks.Each participant will be followed for two months. Their treatment and nurse coaching will also continue for two months. The nurse coach will coach each patient at least four times. Each coaching session will last at least 30 minutes.

   In the evaluation; Dermatological Quality of Life Scale will be used with the global evaluation of the patient and the doctor.

   Approval was obtained from Medipol University Traditional and Alternative Medicine Practices Ethics Committee for the research.
6. Conditions and Keywords Propolis, foot care, nursing education
7. Study Design: Randomised Controlled Trial
8. Arms, Groups, and Interventions There are 2 experiments and 1 control group in the study. Routine antifungal therapy will be applied to all groups. Apart from this, one group will be given propolis, another group will be given plassebo. Another group will be given foot care training.
9. Outcome Measures

   Doctor's global assessment Patient's global assesment Dermatological quality of life scale
10. Eligibility The study was planned in accordance with the Turkish Ministry of Health rules.
11. Contacts, Locations, and Investigator Information Rukiye Burucu Necmettin Erbakan Üniversitesi Seydişehir SBF Seydişehir/ Konya rburucu@hotmail.com 05062347525
12. IPD Sharing Statement...

ELIGIBILITY:
Inclusion Criteria:

* Not being pregnant
* Not being breastfeeding
* Not having confusion
* Not being immunosuppressed
* Not using systemic cortisone
* Not having any dermatological problems (psoriasis, contact dermatitis, etc.) that will affect the treatment.
* Agree to participate in research
* Being accessible by phone
* Having no problems communicating by phone
* Not having problems with physical care

Exclusion Criteria:

* Pregnant / nursing women
* Using systemic antifungal therapy
* Using systemic croticosteroids
* In the process of treatment for oncological reasons
* Are using immunosuppressants
* Dermatological disease (contact dermatitis, psoriasis)
* Under the age of 18 and over the age of 64
* Have cognitive problems
* There is no telephone / telephone number within reach
* Individuals who have difficulties in speaking and understanding Turkish will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Evaluation | 3 month
  Dermatological Quality of Life Scale

SECONDARY OUTCOMES:
Doctor's an patient's global | 3 month
  Doctor's global assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Univercity, Konya, Turkey (Türkiye)